CLINICAL TRIAL: NCT04625907
Title: FaR-RMS: An Overarching Study for Children and Adults With Frontline and Relapsed RhabdoMyoSarcoma
Acronym: FaR-RMS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_17-247; 2018-000515-24 (EudraCT Number); 45535982 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2019-11-22; First posted 2020-11-12 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Irinotecan; Dactinomycin; Doxorubicin; Ifosfamide; Vincristine; Vinorelbine; Cyclophosphamide; Temozolomide; Radiotherapy; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (19):
- Phase 1b Dose finding: VHR induction - IRIVA (Experimental): Irinotecan: an i.v. infusion over 1 hour on days 8,9,10,11 and 12 . For the phase 1b registration, starting dose of 20 mg/m2.
  Ifosfamide: 3g/m2 as an i.v. infusion over 3 hours on days 1 and 2 Vincristine: 1.5 mg/m2 as an As per local practice: recommended as a short infusion (maximum dose 2mg). Administered days 1,8,15 on cycles 1-2 and on days 1 and 8 on cycles 3-9.
  Actinomycin: 1.5 mg/m2 as an i.v. bolus injection (maximum dose 2mg) on day 1.
  Interventions: Drug: Irinotecan; Drug: Actinomycin D; Drug: Ifosfamide; Drug: Vincristine
- CT1A: VHR induction - IVADO (Active Comparator): Ifosfamide: 3g/m2 as an i.v. infusion over 3 hours on days 1 and 2 Vincristine: 1.5 mg/m2 As per local practice: recommended as a short infusion (maximum dose 2mg). Administered days 1,8,15 on cycles 1-2 and on day 1 on cycles 3-9.
  Actinomycin: 1.5 mg/m2 as an i.v. bolus injection (maximum dose 2mg) on day 1. Doxorubicin: 30 mg/m2 as an i.v infusion over 1 hour on days 1 and 2 on cycles 1-4
  Interventions: Drug: Actinomycin D; Drug: Doxorubicin; Drug: Ifosfamide; Drug: Vincristine
- CT1A: VHR Induction IRIVA (Experimental): Irinotecan: an i.v. infusion over 1 hour on days 8,9,10,11 and 12 . Phase 2 recommended dose as determined by IRIVA dose finding arm Ifosfamide: 3g/m2 as an i.v. infusion over 3 hours on days 1 and 2 Vincristine: 1.5 mg/m2 As per local practice: recommended as a short infusion (maximum dose 2mg). Administered days 1,8,15 on cycles 1-2 and on days 1 and 8 on cycles 3-9.
  Actinomycin: 1.5 mg/m2 as an i.v. bolus injection (maximum dose 2mg) on day 1.
  Interventions: Drug: Irinotecan; Drug: Actinomycin D; Drug: Ifosfamide; Drug: Vincristine
- CT1B: HR Induction IVA (Active Comparator): Ifosfamide: 3g/m2 as an i.v. infusion over 3 hours on days 1 and 2 Vincristine: 1.5 mg/m2 As per local practice: recommended as a short infusion (maximum dose 2mg). Administered days 1,8,15 on cycles 1-2 and on day 1 on cycles 3-9.
  Actinomycin: 1.5 mg/m2 as an i.v. bolus injection (maximum dose 2mg) on day 1.
  Interventions: Drug: Actinomycin D; Drug: Ifosfamide; Drug: Vincristine
- CT1B: HR Induction IRIVA (Experimental): Irinotecan: an i.v. infusion over 1 hour on days 8,9,10,11 and 12 . Phase 2 recommended dose as determined by IRIVA dose finding arm Ifosfamide: 3g/m2 as an i.v. infusion over 3 hours on days 1 and 2 Vincristine: 1.5 mg/m2 As per local practice: recommended as a short infusion (maximum dose 2mg). Administered days 1,8,15 on cycles 1-2 and on days 1 and 8 on cycles 3-9.
  Actinomycin: 1.5 mg/m2 as an i.v. bolus injection (maximum dose 2mg) on day 1.
  Interventions: Drug: Irinotecan; Drug: Actinomycin D; Drug: Ifosfamide; Drug: Vincristine
- RT1A: Preoperative Radiotherapy (Experimental): To be given either 41.4 Gy or 50.4 Gy prior to surgery
  Interventions: Radiation: radiotherapy
- RT1A: Post operative radiotherapy (Active Comparator): To be given either 41.4 Gy or 50.4 Gy following surgery
  Interventions: Radiation: radiotherapy
- RT1B: Radiotherapy for resectable disease: dose escalated (Experimental): To receive 50.4 Gy
  Interventions: Radiation: radiotherapy
- RT1B: Radiotherapy for resectable disease: standard dose (Active Comparator): To receive 41.4 Gy
  Interventions: Radiation: radiotherapy
- RT1C: Radiotherapy for unresectable disease: dose escalated (Experimental): To receive 59.4 Gy
  Interventions: Radiation: radiotherapy
- RT1C: Radiotherapy for unresectable disease: standard dose (Active Comparator): To receive 50.4 Gy
  Interventions: Radiation: radiotherapy
- RT2: Radiotherapy to primary tumour and involved lymph nodes (Experimental): Radiotherapy to the primary tumour and involved regional lymph nodes only
  Interventions: Radiation: radiotherapy
- RT2: Radiotherapy to all metastatic sites (Experimental): Radiotherapy given to all metastatic sites
  Interventions: Radiation: radiotherapy
- CT2A: VHR Maintenance - VC (Experimental): Vinorelbine: 25 mg/m2 i.v. or 60 mg/m2 orally on days 1,8 and 15 Cyclophosphamide 25 mg/m2 orally daily for 28 days
  Interventions: Drug: Vinorelbine; Drug: Cyclophosphamide
- CT2A: Maintenance -Stop treatment (No Intervention): To stop treatment at the point of randomisation
- CT2B: HR Maintenance - VC (Experimental): Vinorelbine: 25 mg/m2 i.v. on days 1,8 and 15 Cyclophosphamide 25 mg/m2 orally daily for 28 days
  Interventions: Drug: Vinorelbine; Drug: Cyclophosphamide
- CT2B: HR Maintenance - Stop Treatment (No Intervention): To stop treatment at the point of randomisation
- CT3: Relpased Chemotherapy - VIRT (Active Comparator): Vincristine: 1.5 mg/m2 As per local practice: recommended as a short infusion (maximum dose 2mg) on days 1 and 8 Irinotecan: 50 mg/m2 as an i.v. infusion over 1 hour on days 1-5 Temozolomide: 125 mg/m2 (Escalate to 150mg/m2/day in Cycle 2 if no toxicity > grade 3) as an oral tablets prior to vincristine and irinotecan on days 1-5
  Interventions: Drug: Irinotecan; Drug: Vincristine; Drug: Temozolomide
- CT3: Relapsed Chemotherapy - VIRR (Experimental): Vincristine: 1.5 mg/m2 As per local practice: recommended as a short infusion (maximum dose 2mg) on days 1 and 8 Irinotecan: 50 mg/m2 as an i.v. infusion over 1 hour on days 1-5 Regorafenib: Children between 6 and 24 months = 65 mg/m2, children less than 12 and/or less than 40kg dose = 82 mg/m2 Maximum 120 mg, Fixed dose of 120 mg for patients over 12 years of age AND ≥ 40 kg, as an oral tablets on days 8 to 21.
  Interventions: Drug: Irinotecan; Drug: Vincristine; Drug: Regorafenib

INTERVENTIONS:
Drug: Irinotecan — antineoplastic enzyme inhibitor
  Arms: CT1A: VHR Induction IRIVA; CT1B: HR Induction IRIVA; CT3: Relapsed Chemotherapy - VIRR; CT3: Relpased Chemotherapy - VIRT; Phase 1b Dose finding: VHR induction - IRIVA
Drug: Actinomycin D — Antineoplastic agent that is a polypeptide antibiotic
  Other Names: Dactinomycin
  Arms: CT1A: VHR Induction IRIVA; CT1A: VHR induction - IVADO; CT1B: HR Induction IRIVA; CT1B: HR Induction IVA; Phase 1b Dose finding: VHR induction - IRIVA
Drug: Doxorubicin — An anthracycline topoisomerase inhibitor isolated from streptpmyces peucetius var. casesius
  Arms: CT1A: VHR induction - IVADO
Drug: Ifosfamide — chemotherapeutic agent chemically related to the nitrogen mustards and is a synthetic analog of cyclophosphamide
  Arms: CT1A: VHR Induction IRIVA; CT1A: VHR induction - IVADO; CT1B: HR Induction IRIVA; CT1B: HR Induction IVA; Phase 1b Dose finding: VHR induction - IRIVA
Drug: Vincristine — anti neoplastic vinca alkaloid agent
  Arms: CT1A: VHR Induction IRIVA; CT1A: VHR induction - IVADO; CT1B: HR Induction IRIVA; CT1B: HR Induction IVA; CT3: Relapsed Chemotherapy - VIRR; CT3: Relpased Chemotherapy - VIRT; Phase 1b Dose finding: VHR induction - IRIVA
Drug: Vinorelbine — vinca alkaloid with a role as an antineoplastic agent
  Arms: CT2A: VHR Maintenance - VC; CT2B: HR Maintenance - VC
Drug: Cyclophosphamide — Precursor of an alkylating nitrogen mustard antineoplastic and immunosuppressive agent
  Arms: CT2A: VHR Maintenance - VC; CT2B: HR Maintenance - VC
Drug: Temozolomide — oral antineoplastic alkylating agent
  Arms: CT3: Relpased Chemotherapy - VIRT
Radiation: radiotherapy — Ionising radiation
  Arms: RT1A: Post operative radiotherapy; RT1A: Preoperative Radiotherapy; RT1B: Radiotherapy for resectable disease: dose escalated; RT1B: Radiotherapy for resectable disease: standard dose; RT1C: Radiotherapy for unresectable disease: dose escalated; RT1C: Radiotherapy for unresectable disease: standard dose; RT2: Radiotherapy to all metastatic sites; RT2: Radiotherapy to primary tumour and involved lymph nodes
Drug: Regorafenib — Oral multi-kinase inhibitor that targets a broad range of angiogenic, stromal and oncogenic kinases, including vascular endothelial growth factor receptors (VEFGR) 1, 2 and 3, tyrosine kinase with immunoglobulin and epidermal growth factor homology domain 2 (TIE2), platelet-derived growth factor receptor (PDGFR), fibroblast growth factor receptors (FGFR), c-KIT, RET, RAF-1 and BRAF (wild-type and V600E mutant).
  Arms: CT3: Relapsed Chemotherapy - VIRR

SUMMARY:
FaR-RMS is an over-arching study for children and adults with newly diagnosed and relapsed rhabdomyosarcoma (RMS)

DETAILED DESCRIPTION:
FaR-RMS is an over-arching study for children and adults with newly diagnosed and relapsed rhabdomyosarcoma (RMS). It is a multi-arm, multi-stage format, involving several different trial questions. FaR-RMS is intended to be a rolling programme of research with new treatment arms being introduced dependant on emerging data and innovation. This study has multiple aims. It aims to evaluate the impact of new agent regimens in both newly diagnosed and relapsed RMS; whether changing the duration of maintenance therapy affects outcome; and whether changes to dose, extent (in metastatic disease) and timing of radiotherapy improve outcome and quality of life. In addition the study will evaluate risk stratification through the use of PAX-FOXO1 fusion gene status instead of histological subtyping and explore the use of FDG PET-CT response assessment as a prognostic biomarker for outcome following induction chemotherapy.

Newly diagnosed patients should, where possible, be entered into the FaR-RMS study at the time of first diagnosis prior to receiving any chemotherapy. However, patients can enter at the point of radiotherapy or maintenance, and those with relapsed disease can enter the study even if not previously entered at initial diagnosis. Patients may be entered into more than one randomisation/registration, dependant on patient risk group and disease status.

ELIGIBILITY:
Inclusion Criteria for study entry - Mandatory at first point of study entry

1. Histologically confirmed diagnosis of RMS (except pleomorphic RMS)
2. Written informed consent from the patient and/or the parent/legal guardian

Phase 1b Dose Finding - IRIVA Inclusion

1. Entered in to the FaR-RMS study at diagnosis
2. Very High Risk disease
3. Age >12 months and ≤25 years
4. No prior treatment for RMS other than surgery
5. Medically fit to receive treatment
6. Adequate hepatic function:

   1. Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age, unless the patient is known to have Gilbert's syndrome
   2. ALT or AST < 2.5 X ULN for age
7. Absolute neutrophil count ≥1.0x 109/L
8. Platelets ≥ 80 x 109/L
9. Adequate renal function: estimated or measured creatinine clearance ≥60 ml/min/1.73 m2
10. Documented negative pregnancy test for female patients of childbearing potential
11. Patient agrees to use contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where patient is sexually active
12. Written informed consent from the patient and/or the parent/legal guardian

Exclusion

1. Weight <10kg
2. Active > grade 2 diarrhoea
3. Prior allo- or autologous Stem Cell Transplant
4. Uncontrolled inter-current illness or active infection
5. Pre-existing medical condition precluding treatment
6. Urinary outflow obstruction that cannot be relieved prior to starting treatment
7. Active inflammation of the urinary bladder (cystitis)
8. Known hypersensitivity to any of the treatments or excipients
9. Second malignancy
10. Pregnant or breastfeeding women

Frontline chemotherapy randomisation Very High Risk - CT1a Inclusion

1. Entered in to the FaR-RMS study at diagnosis
2. Very High Risk disease
3. Age ≥ 6 months
4. Available for randomisation ≤60 days after diagnostic biopsy/surgery
5. No prior treatment for RMS other than surgery
6. Medically fit to receive treatment
7. Adequate hepatic function :

   a. Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age, unless the patient is known to have Gilbert's syndrome
8. Absolute neutrophil count ≥1.0x 109/L (except in patients with documented bone marrow disease)
9. Platelets ≥ 80 x 109/L (except in patients with documented bone marrow disease)
10. Fractional Shortening ≥ 28%
11. Documented negative pregnancy test for female patients of childbearing potential
12. Patient agrees to use contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where patient is sexually active
13. Written informed consent from the patient and/or the parent/legal guardian

Exclusion

1. Active > grade 2 diarrhoea
2. Prior allo- or autologous Stem Cell Transplant
3. Uncontrolled inter-current illness or active infection
4. Pre-existing medical condition precluding treatment
5. Urinary outflow obstruction that cannot be relieved prior to starting treatment
6. Active inflammation of the urinary bladder (cystitis)
7. Known hypersensitivity to any of the treatments or excipients
8. Second malignancy
9. Pregnant or breastfeeding women

Frontline chemotherapy randomisation High Risk - CT1b Inclusion

1. Entered in to the FaR-RMS study at diagnosis
2. High Risk disease
3. Age ≥ 6 months
4. Available for randomisation ≤60 days after diagnostic biopsy/surgery
5. No prior treatment for RMS other than surgery
6. Medically fit to receive treatment
7. Adequate hepatic function :

   a. Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age, except if the patient is known to have Gilbert's syndrome
8. Absolute neutrophil count ≥1.0x 109/L
9. Platelets ≥ 80 x 109/L
10. Documented negative pregnancy test for female patients of childbearing potential
11. Patient agrees to use contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where patient is sexually active
12. Written informed consent from the patient and/or the parent/legal guardian

Exclusion

1. Active > grade 2 diarrhoea
2. Prior allo- or autologous Stem Cell Transplant
3. Uncontrolled inter-current illness or active infection
4. Pre-existing medical condition precluding treatment
5. Urinary outflow obstruction that cannot be relieved prior to starting treatment
6. Active inflammation of the urinary bladder (cystitis)
7. Known hypersensitivity to any of the treatments or excipients
8. Second malignancy
9. Pregnant or breastfeeding women

Frontline Radiotherapy Note: eligible patients may enter multiple radiotherapy randomisations.

Radiotherapy Inclusion - for all radiotherapy randomisations

1. Entered in to the FaR-RMS study (at diagnosis or prior to radiotherapy randomisation)
2. Very High Risk, High Risk and Standard Risk disease
3. ≥ 2 years of age
4. Receiving frontline induction treatment as part of the FaR-RMS trial or with a IVA/IVADo based chemotherapy regimen patients for whom. Note that patients for whom ifosfamide has been replaced with cyclophosphamide will be eligible
5. Patient assessed as medically fit to receive the radiotherapy
6. Documented negative pregnancy test for female patients of childbearing potential
7. Patient agrees to use contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where patient is sexually active
8. Written informed consent from the patient and/or the parent/legal guardian

Radiotherapy Exclusion - for all radiotherapy randomisations

1. Prior allo- or autologous Stem Cell Transplant
2. Second malignancy
3. Pregnant or breastfeeding women
4. Receiving radiotherapy as brachytherapy

RT1a Specific Inclusion

1. Primary tumour deemed resectable (predicted R0/ R1 resection feasible) after 3 cycles of induction chemotherapy (6 cycles for metastatic disease)
2. Adjuvant radiotherapy required in addition to surgical resection (local decision).
3. Available for randomisation after cycle 3 and prior to the start of cycle 6 of induction chemotherapy for localised disease, or after cycle 6 and prior to the start of cycle 9 for metastatic disease

RT1b Specific Inclusion

1. Primary tumour deemed resectable (predicted R0/R1 resection) after 3 cycles of induction chemotherapy (6 cycles for metastatic disease).
2. Adjuvant radiotherapy required in addition to surgical resection (local decision)
3. Higher Local Failure Risk (HLFR) based on presence of either of the following criteria:

   1. Unfavourable site
   2. Age ≥ 18yrs
4. Available for randomisation after cycle 3 and prior to the start of cycle 6 of induction chemotherapy for localised disease, or after cycle 6 and prior to the start of cycle 9 for metastatic disease

RT1c Specific Inclusion

1. Primary radiotherapy indicated (local decision)
2. Higher Local Failure Risk (HLFR) based on either of the following criteria:

   1. Unfavourable site
   2. Age ≥ 18yrs
3. Available for randomisation after cycle 3 and prior to the start of cycle 6 of induction chemotherapy for localised disease, or after cycle 6 and prior to the start of cycle 9 for metastatic disease

RT2

1. Available for randomisation after cycle 6 and before the start of cycle 9 of induction chemotherapy.
2. Unfavourable metastatic disease, defined as Modified Oberlin Prognostic Score 2-4

   * Note: Definition of metastatic lesions for RT2 eligibility

Modified Oberlin Prognostic Score (1 point for each adverse factor):

* Age ≥10y
* Extremity, Other, Unidentified Primary Site
* Bone and/ or Bone Marrow involvement
* ≥3 metastatic sites

Unfavourable metastatic disease: 2- 4 adverse factors Favourable metastatic disease: 0-1 adverse factors

Maintenance chemotherapy (Very High Risk) - CT2a Inclusion Randomisation must take place during the 12th cycle of maintenance chemotherapy.

1. Entered in to the FaR-RMS study (at diagnosis or at any subsequent time point)
2. Very High Risk disease
3. Received frontline induction chemotherapy as part of the FaR-RMS trial or with a IVA/IVADo based chemotherapy regimen

   a. Patients for whom ifosfamide has been replaced with cyclophosphamide will be eligible
4. Completed 11 cycles of VnC maintenance treatment (either oral or IV regimens)
5. No evidence of progressive disease
6. Absence of severe vincristine neuropathy - i.e requiring discontinuation of vincristine treatment)
7. Medically fit to continue to receive treatment
8. Patient agrees to use contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where patient is sexually active
9. Written informed consent from the patient and/or the parent/legal guardian

Exclusion

1. Prior allo- or autologous Stem Cell Transplant
2. Uncontrolled intercurrent illness or active infection
3. Urinary outflow obstruction that cannot be relieved prior to starting treatment
4. Active inflammation of the urinary bladder (cystitis)
5. Second malignancy
6. Pregnant or breastfeeding women

Maintenance chemotherapy (High Risk) - CT2b Randomisation must take place during the 6th cycle of maintenance chemotherapy. Inclusion

1. Entered in to the FaR-RMS study (at diagnosis or at any subsequent time point)
2. High Risk disease
3. Received frontline induction chemotherapy as part of the FaR-RMS trial or with a IVA based chemotherapy regimen. Note that patients for whom ifosfamide has been replaced with cyclophosphamide will be eligible
4. Completed 5 cycles of VnC maintenance treatment
5. No evidence of progressive disease
6. Absence of severe vincristine neuropathy i.e. requiring discontinuation of vincristine treatment
7. Medically fit to continue to receive treatment
8. Patient agrees to use contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where patient is sexually active
9. Written informed consent from the patient and/or the parent/legal guardian

Exclusion

1. Prior allo- or autologous Stem Cell Transplant
2. Uncontrolled inter current illness or active infection
3. Urinary outflow obstruction that cannot be relieved prior to starting treatment
4. Active inflammation of the urinary bladder (cystitis)
5. Second malignancy
6. Pregnant or breastfeeding women

CT3 Relapsed Chemotherapy

Inclusion:

1. Entered in to the FaR-RMS study (at diagnosis or at any subsequent time point)
2. First or subsequent relapse of histologically verified RMS
3. Age ≥ 6 months
4. Measurable or evaluable disease
5. No cytotoxic chemotherapy or other investigational medicinal product (IMP) within previous three weeks: within two weeks for vinorelbine and cyclophosphamide maintenance chemotherapy
6. Medically fit to receive trial treatment
7. Documented negative pregnancy test for female patients of childbearing potential within 7 days of planned randomisation
8. Patient agrees to use contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where patient is sexually active
9. Written informed consent from the patient and/or the parent/legal guardian

Exclusion:

1. Progression during frontline therapy without previous response (=Refractory to first line treatment)
2. Prior regorafenib or temozolomide
3. Active > grade 1 diarrhoea
4. ALT or AST >3.0 x upper limit normal (ULN)
5. Bilirubin, Total >1.5 x ULN; total bilirubin is allowed up to 3 x ULN if Gilbert's syndrome is documented
6. Patients with unstable angina or new onset angina (within 3 months of planned date of randomisation), recent myocardial infarction (within 6 months of randomisation) and those with cardiac failure New York Heart Association (NYHA) Classification 2 or higher Cardiac abnormalities such as congestive heart failure (Modified Ross Heart Failure Classification for Children = class 2) and cardiac arrhythmias requiring antiarrhythmic therapy (beta blockers or digoxin are permitted)
7. Uncontrolled hypertension > 95th centile for age and gender
8. Prior allo- or autologous Stem Cell Transplant
9. Uncontrolled inter-current illness or active infection
10. Pre-existing medical condition precluding treatment
11. Known hypersensitivity to any of the treatments or excipients
12. Second malignancy
13. Pregnant or breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1672 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (RT2) | From randomisation to first failure event, timeframe 36 months
  Failure events are:
  * Relapse or progression of existing disease, or occurrence of disease at new sites,
  * Death from any cause without disease progression,
  * Second malignant neoplasm
Event Free Survival (CT1A) | From randomisation to first failure event, timeframe 36 months
  Failure events are:
  * Relapse or progression of existing disease, or occurrence of disease at new sites,
  * Death from any cause without disease progression,
  * Second malignant neoplasm
Event Free Survival (CT1B) | From randomisation to first failure event, timeframe 36 months
  Failure events are:
  * Relapse or progression of existing disease, or occurrence of disease at new sites,
  * Death from any cause without disease progression,
  * Second malignant neoplasm
Event Free Survival (CT2A) | From randomisation to first failure event, timeframe 36 months
  Failure events are:
  * Relapse or progression of existing disease, or occurrence of disease at new sites,
  * Death from any cause without disease progression,
  * Second malignant neoplasm
Event Free Survival (CT2B) | Time from randomisation to first failure event, timeframe 36 months
  Failure events are:
  * Relapse or progression of existing disease, or occurrence of disease at new sites,
  * Death from any cause without disease progression,
  * Second malignant neoplasm
Event Free Survival (CT3) | Patients will be followed up for a minimum of 6 years from trial entry (or 5 years from end of relapsed trial treatment, whichever comes later). Patients will be followed up for progression and death until the end of trial definition has been met.
  To determine whether new systemic therapy regimens improve event free survival in relapsed RMS compared to standard therapy (VIRT) (CT3):
  Initial new systemic therapy combination to be tested:
  o Regorafenib (R) added to vincristine and irinotecan (VIR) (VIRR)
Local Failure Free Survival (RT1A and RT1B) | Time from randomisation to first local failure event, timeframe 36 months
  A local failure event is relapse or progression of tumour at the primary site at any time even if there has been a prior /concurrent, regional or distant failure
Local Failure Free Survival (RT1C) | Time from randomisation to first local failure event, timeframe 36 months
  A local failure event is relapse or progression of tumour at the primary site at any time even if there has been a prior /concurrent, regional or distant failure

SECONDARY OUTCOMES:
Recommended Phase II Dose (Phase 1b) | From first patient first visit in dose finding study until appropriate dose level found, estimated 9 months
  Based on tolerability, where tolerability is evaluated through the occurrence of dose limiting toxicity (DLT).
Maximum Tolerated Dose (Phase 1b) | From first patient first visit in dose finding study until appropriate dose level
  Dose level at which no or one participant experiences a DLT when at least two of three to six participants experience a DLT at the next highest dose.
Toxicity (All chemotherapy randomisations) | From date of protocol defined treatment until 30 days after the administration of the last treatment
  Categorised and graded using Common Terminology Criteria for Adverse Events
Dose Limiting Toxicity (Phase 1b) | From commencement of treatment until 21 days after the start of cycle 2 (each cycle is 21 days)
  Diarrhoea: Grade 3 for >3 days despite loperamide therapy Diarrhoea: Grade 4 despite loperamide therapy. Enterocolitis: Grade 3 or above Ileus: Grade 3 or above for more than 3 days Oral mucositis: Grade 3 above for >3 days despite optimal supportive care Persistent neutropenia or thrombocytopenia leading to delay of start of next course by >7 days; i.e. starting > day 28 Any grade 3 or 4 toxicity resulting in discontinuation of the new combination Any grade 5 toxicity
Response (Phase 1b, CT1A, CT1B) | Response assessed after course 3 (63 days) and 6 (126 days)
  defined as complete (CR) or partial response (PR) and is clinically defined. Patients who are not assessable for response - e.g. because of early stopping of treatment or death - will be assumed to be non-responders.
Tolerability (CT3) | From registration/randomisation until death/study endpoint
  To determine the tolerability of the regimens.
Overall Survival (CT1A) | From randomisation to death from any cause, assessed for 36 months
  Death from any cause
Overall Survival (CT1B) | From randomisation to death from any cause, assessed for 36 months
  Death from any cause
Overall Survival (CT2A) | From randomisation to death from any cause, assessed for 36 months
  Death from any cause
Overall Survival (CT2B) | From randomisation to death from any cause, assessed for 36 months
  Death from any cause
Overall Survival (RT1A and RT1B) | From randomisation to death from any cause, assessed for 36 months
  Death from any cause
Overall Survival (RT1C) | From RT1C randomisation to death from any cause, assessed for 36 months
  Death from any cause
Overall Survival (RT2) | From RT2 randomisation to death from any cause, as assessed for 36 months
  Death from any cause
Overall Survival (CT3) | Patients will be followed up for a minimum of 6 years from trial entry (or 5 years from end of relapsed trial treatment, whichever comes later). Patients will be followed up for progression and death until the end of trial definition has been met.
  To evaluate the anti-tumour activity and effect on overall survival of VIRR when compared to standard therapy
Overall Survival (all patients) | From randomisation/registration to death from any cause, assessed for 36 months
  Death from any cause
Acute wound complications and post-operative complications (RT1A and RT1B) | Within 120 days from surgery
  specific grade 3 and above complications according to CTCAE v 4 and Clavien Dindo scale. Specific wound complications within the same time frame will also be collected
Acute post-radiotherapy complications (All radiotherapy randomisations) | Within 120 days from start of radiotherapy
  any grade 3 and above event according to CTCAE v 4
Late complications (RT1A, RT1B. RT1C) | After 120 days from last local therapy
  specific grade 3 and above events according to CTCAE and Clavien-Dindo scale
Loco-regional failure-free survival (All radiotherapy randomisations) | From randomisation to first local and/or regional failure event, assessed for 36 months
  A local failure event is relapse or progression of tumour at the primary site at any time even if there has been a prior concurrent local, regional or distant failure. A regional event is relapse or progression of tumour at regional lymph nodes at any time even if there has been a prior distant failure.
Health related quality of life (RT1A and RT2) self-reported questionnaire completed by patient | 4 timepoints: 1) 1 day of start of radiotherapy, 2) at completion of radiotherapy, average 5 weeks after start of radiotherapy, 3) 3 months and 4) 24 months following radiotherapy
  will be assessed using Pediatric quality of life questionnaire (PedsQL) for the paediatric population (under 18 years). The minimum score is 0 where quality of life is completely unaffected by the intervention to 4 where quality of life is severely affected.
Health related quality of life (RT1A and RT2) self-reported questionnaire completed by the patient | 4 timepoints: 1) 1 day of start of radiotherapy, 2) at completion of radiotherapy, average 5 weeks after start of radiotherapy, 3) 3 months and 4) 24 months following radiotherapy
  will be assessed using European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire 30 (EORTC QLQ-C30) for patients 18 years of age and over. The minimum score is 0 where quality of life is completely unaffected by the intervention to 4 where quality of life is severely affected.
Health related quality of life (CT3) self-reported questionnaire completed by the patient | 3 timepoints: Each Cycle is 28 days. Timepoint 1: Day 0 of cycle 1 (prior to starting treatment), Timepoint 2 day 0 cycle 3, Timepoint 3) day 0 cycle 5
  will be assessed using Pediatric quality of life questionnaire (PedsQL) for the paediatric population (under 18 years). The minimum score is 0 where quality of life is completely unaffected by the intervention to 4 where quality of life is severely affected.
Health related quality of life (CT3) self-reported questionnaire completed by the patient | 3 timepoints: Each Cycle is 28 days. Timepoint 1: Day 0 of cycle 1 (prior to starting treatment), Timepoint 2 day 0 cycle 3, Timepoint 3) day 0 cycle 5
  will be assessed using European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire 30 (EORTC QLQ-C30) for patients 18 years of age and over. The minimum score is 0 where quality of life is completely unaffected by the intervention to 4 where quality of life is severely affected.
Acceptability and Palatability of Regorafenib (CT3) | 1 timepoint: Day 8 of cycle 1 (Each Cycle is 28 days)
  "Acceptability and Palatability Questionnaire" To evaluate the acceptability and palatability of regorafenib formulations
PET Response (if participating in PET Sub-study) | After three cycles of chemotherapy (each cycle is 21 days)
  assessed by PERCIST criteria and visual 'Deauville like' criteria
Event Free Survival (all patients) | From date of randomisation/registration to death from any cause, assessed for 36 months
  Failure events are:
  * Relapse or progression of existing disease, or occurrence of disease at new sites,
  * Death from any cause without disease progression,
  * Second malignant neoplasm
Event Free Survival (if participating in PET Sub-study) | From date of randomisation/registration to death from any cause, assessed for 36 months
  Failure events are:
  * Relapse or progression of existing disease, or occurrence of disease at new sites,
  * Death from any cause without disease progression,
  * Second malignant neoplasm
Local Failure Free Survival (if participating in PET Sub-study) | From date of randomisation/registration to first local failure event, assessed for 36 months
  A local failure event is relapse or progression of tumour at the primary site at any time even if there has been a prior /concurrent, regional or distant failure

CONTACTS AND LOCATIONS:
Overall Officials: Meriel Jenney, Principal Investigator — Chief Investigator
Locations (128):
- Australia (11):
  - Queensland Children's Hospital, Brisbane
  - Chris O'brien Lifehouse, Camperdown
  - Monash Children's Hospital, Clayton
  - Peter Maccallum Cancer Centre, Melbourne
  - Royal Childrens Hospital Melbourne, Melbourne
  - John Hunter Children's Hospital, New Lambton Heights
  - Perth Children's Hospital, Perth
  - Sydney Children's Hospital, Sydney
  - The Childrens Hospital At Westmead, Sydney
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - Kepler University Clinic Linz, Linz
  - St Anna Childrens Hospital, Vienna
- Belgium (6):
  - Cliniques Universitaires Saint Luc, Brussels
  - Hopital Universitaire Des Enfants Reine Fabiola, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Uz Leuven Campus Gasthuisberg, Leuven
  - Centre Hospitalier Regional De La Citadelle, Liège
  - Clinique Chc Montlegia, Liège
- Masaryk University Hospital Brno, Brno, Czechia
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - University Hospital Rigshospitalet, Copenhagen
- France (27):
  - Centre Hospitalier Universitaire D'angers, Angers
  - Centre Hospitalier Regional Universitaire Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire De Bordeaux - Hopital Pellegrin, Bordeaux
  - Centre Hospitalier Regional Universitaire Brest - Hopital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Universitaire De Caen, Caen
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hopital D'enfants, Dijon
  - Centre Hospitalier Universitaire De Grenoble, Grenoble
  - Centre Hospitalier Universitaire La Reunion, La Réunion
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital De La Timone (ap-hm), Marseille
  - Centre Hospitalier Universitaire De Nancy, Nancy
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Hopital Armand Trousseau, Paris
  - Institut Curie, Paris
  - Centre Hospitalier Universitaire Haut Levque, Pessac
  - Centre Hospitalier Universitaire De Poitiers, Poitiers
  - Chu De Reims, Reims
  - Centre Eugne Marquis De Rennes, Rennes
  - Centre Hospitalier Universitaire De Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire De Rouen, Rouen
  - Centre Hospitalier Universitaire Saint-etienne, Saint-Etienne
  - Strasbourg Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire De Toulouse - Hopital Des Enfants, Toulouse
  - Centre Hospitalier Regional Universitaire De Tours - Hopital Clocheville, Tours
  - Gustave Roussy, Villejuif
- Greece (8):
  - Children's General Hospital P and A Kyriakou, Athens
  - Department of Pediatric Hematology-oncology - Aghia Sophia Children's Hospital, Athens
  - Hellenic Society of Pediatric Hematology- Oncology, Athens
  - University Unit of Pediatric Oncology-hematology - Children's Hospital Agia Sophia, Athens
  - Children's and Adolescent's Oncology Clinic, "MITERA" Children's Hospital, Attiki
  - Hematology-oncology Children's Clinic, University General Hospital of Heraklion, Heraklion
  - Ahepa University General Hospital of Thessaloniki, Thessaloniki
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Our Lady's Children's Hospital, Crumlin, Ireland
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Medical Centre, Jerusalem
  - Schneider Medical Centre, Petah Tikva
  - Dana Children's Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Centre, Tel Litwinsky
- University Hospital of Padova (azienda Ospedaliera of Padua), Padua, Italy
- Netherlands (2):
  - University Medical Centre Groningen, Groningen
  - Prinses Maxima Centrum Voor Kinderoncologie, Utrecht
- New Zealand (2):
  - Starship Children's Health, Auckland
  - Christchurch Hospital, Christchurch
- Norway (5):
  - Haukeland University Hospital - Paediatric, Bergen
  - Oslo University Hospital - Paediatrics, Oslo
  - Oslo University Hospital - Radiumhospitalet, Oslo
  - University Hospital of North Norway - Paediatric, Tromsø
  - St Olavs Hospital - Paediatric, Trondheim
- Instituto Portugues De Oncologia De Losbona Francisco Gentil, Epe, Lisbon, Portugal
- Bratislava, National Institute for Children's Diseases, Bratislava, Slovakia
- Slovenia (2):
  - University Childrens Hospital Ljubljana, Ljubljana
  - University Medical Centre Ljubjlana, Ljubljana
- Spain (10):
  - Hospital Sant Joan De Deu, Barcelona
  - Hospital Universitari Vall D'hebron, Barcelona
  - Hospital De Cruces, Bilbao
  - Hospital Del Nino Jesus, Madrid
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario De Malaga, Málaga
  - Hospital Virgen Del Rocio, Seville
  - Hospital Politecnico U La Fe, Valencia
  - Hospital Universitario Miguel Servet Materno - infantil, Zaragoza
- Uppsala University Childrens Hospital, Uppsala, Sweden
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitats-kinderspital Bieder Basel (UKBB), Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Hug Hopitaux Universitaires De Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Lausanne
  - Luzerner Kantonspital - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - Universitaetsspital Zurich, Zurich
- United Kingdom (31):
  - Royal Marsden Hospital, Sutton, Surrey
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Belfast City Hospital, Belfast
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - The Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology And Oncology Centre, Bristol
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Noah's Ark Children's Hospital for Wales, Cardiff
  - Velindre Hospital, Cardiff
  - Royal Hospital for Children and Young People, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Hospital for Children Glasgow, Glasgow
  - Leeds General Infirmary, Leeds
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital for Children, London
  - Royal Marsden Hospital London, London
  - University College London Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Queen's Medical Centre, Nottingham, Nottingham
  - John Radcliffe Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton